CLINICAL TRIAL: NCT05754294
Title: Electric Polarization of Red Blood Cells "Polaris": A Cohort Study to Assess the Erythrocytes Membrane Integrity Through Charge Conservation, Following Conventional and Minimally Invasive Cardiac Surgery Procedures and The Related Perfusion Techniques
Brief Title: Electric Polarization of Red Blood Cells : A Cohort Study to Assess the Erythrocytes Membrane Integrity Through Charge Conservation, Following Cardiac Surgery.
Acronym: Polaris
Status: Withdrawn | Type: Observational
Why Stopped: absence of funding
Sponsor: Anthea Hospital Bari (Other)
Responsible Party: Principal Investigator, Ignazio Condello, Principal Investigator, Anthea Hospital Bari
Other Study IDs: AntheaH
Record Dates: First submitted 2023-02-22; First posted 2023-03-03 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Inflammatory Response; Erythrocyte Destruction; Red Blood Cell Disorder; Hemolysis; Cardiovascular Disorder
MeSH Terms: conditions — Hemolysis; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Coronary arteries bypass grafting with conventional cardiopulmonary bypass (cCPB): (n=20) patients, were allocated for Conventional Cardiopulmonary Bypass (cCPB)
  Interventions: Diagnostic Test: Polarization of red blood cells
- Coronary arteries bypass grafting with Minimally invasive extracorporeal circulation (MiECC): (n=20) patients, were allocated for Minimal invasive Extracorporeal Circulation (MiECC) type III.
  Interventions: Diagnostic Test: Polarization of red blood cells
- Minimally invasive mitral valve repair (MIMVR) with CPB time (< 60 min.): (n=20) patients, were allocated for Minimally invasive mitral valve repair (MIMVR) with CPB time (< 60 min.)
  Interventions: Diagnostic Test: Polarization of red blood cells
- Minimally invasive mitral valve repair (MIMVR) with CPB time (>100 min.): n=20) patients, were allocated for Minimally invasive mitral valve repair (MIMVR) with CPB time (> 100 min.)
  Interventions: Diagnostic Test: Polarization of red blood cells

INTERVENTIONS:
Diagnostic Test: Polarization of red blood cells — Pre and perioperative data blood sample were collected for each patient 5 minutes (min) before the CPB start and 5 minutes before the end of the CPB for Complete Blood Count (CBC), Erythrocyte Sedimentation Rate (ESR) and Plasma Free Hemoglobin (pFHb). At the end of CPB the residual blood from the extracorporeal circulation was treated with cell-saver and the treated and concentrated red blood cells were collected in a transfusion bag. Two milliliters (ml) was taken from the bag, one ml was subjected to a blood gas test for the evaluation of the Hemoglobin (Hb) content and one ml was subjected inside a cuvette to the release of positive ions (polarization) with a charge of 50 Millivolt (mV) for a time of 5 seconds through charge circuit, after the trend of the conserved charge was measured through a multimeter, instrument that can measure multiple electrical properties.

SUMMARY:
An immediate perioperative parameter that assess the integrity of the Erythrocytes Membrane and therefore their structural quality isn't available in clinical practice and medical diagnostics except through indirect clinical biochemical tests or through the scanning electron microscope. The red blood cell (RBC) membrane contains proteins and glycoproteins embedded in a fluid lipid bilayer that confers viscoelastic behavior. Sialylated glycoproteins of the RBC membrane are responsible for a negatively charged surface which creates a repulsive electric zeta potential (ζ) between cells. These charges help prevent the interaction between RBCs and the other cells and especially between each other. The zeta potential is a physical property which is exhibited by all particles in suspension. The development of a net charge on any particle affects the distribution of ions in the surrounding interfacial region resulting in an increased concentration of counter ions of opposite charge to that of the particle, close to the surface. In this context we present a new parameter that studies the interactions of the Erythrocytes membrane treated with positive ions and their maintenance of the charge. We compared the measured polarization values with the Erythrocyte Sedimentation Rate (ESR), expression of speed with which RBCs tend to settle inside a particular graduated capillary called Westergren's tube and Plasma Free Hemoglobin (pFHb).

ELIGIBILITY:
Inclusion Criteria:

* Elective, primary cardiac surgery
* Minimally invasive cardiac surgery
* Mitral Valve Surgery (MVS)
* Conventional cardiac surgery (CCS)
* Coronary Arterial Bypass Grafting (CABG).

Exclusion Criteria:

* Abnormal plasma lactate levels (>2 mmol/L)
* Renal
* Liver failure,
* Obesity,
* Uncompensated diabetes,
* Autoimmune disease, active infection
* Immunosuppressant therapy
* Coagulation disorder
* Surgery with circulatory arrest
* Preoperative hematocrit (Hct) <27%

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Have been collected a perspective cohort of Eighty elective Cardiac Surgery procedures with Cardiopulmonary bypass (CPB) in a single tertiary institution Anthea Hospital Gvm Care & Research, Bari, Italy. Forty patients were treated for Coronary Artery Bypass Grafting (CABG) of which (n=20), were allocated for Conventional Cardiopulmonary Bypass (cCPB) and (n=20), were allocated for Minimal invasive Extracorporeal Circulation (MiECC) type III. Forty patients were treated for Minimally Invasive Mitral Valve Repair (MIMVR); (n=20), reported a CPB time (< 60 min.) and (n=20), a CPB time (>100 min.).
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Erythrocytes Membrane Integrity | At the end of Cardiopulmonary Bypass
  Conservation of charge after polarization
Erythrocyte Sedimentation Rate (ESR) | At the end of Cardiopulmonary Bypass
  Inflammation
Plasma Free Hemoglobin (pFHb) | At the end of Cardiopulmonary Bypass
  Hemolysis

CONTACTS AND LOCATIONS:
Locations (1):
- Anthea Hospital, Bari, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol